CLINICAL TRIAL: NCT02372669
Title: Chitosan Nerv Tube for Primary Repair of Traumatic Sensory Nerve Lesions of the Hand - a Clinical Randomized Controlled Multicenter Trial
Brief Title: Chitosan Nerv Tube for Primary Repair of Traumatic Sensory Nerve Lesions of the Hand
Acronym: CNT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: BG Unfallklinik Murnau (Other)
Responsible Party: Principal Investigator, Florian Neubrech, MD, BG Unfallklinik Murnau
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BGU-LU-123
Record Dates: First submitted 2015-02-15; First posted 2015-02-26 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Traumatic Lesion of Sensory Nerves of the Hand

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chitosan (Experimental): Enrolled participants presenting with traumatic sensory nerve lesions of the hand without defect zone that were randomized to primary microsurgical repair with the additional use of a chitosan nerve tube.
  Interventions: Device: Chitosan nerve tube in addition to gold standard therapy; Procedure: Gold standard Primary microsurgical repair
- Gold standard alone (Active Comparator): Enrolled participants presenting with traumatic sensory nerve lesions of the hand without defect zone that were randomized to primary microsurgical repair without the additional use of a chitosan nerve tube.
  Interventions: Procedure: Gold standard Primary microsurgical repair

INTERVENTIONS:
Device: Chitosan nerve tube in addition to gold standard therapy — Primary microsurgical repair of traumatic lesion of sensory nerves of the hand with use of an chitosan nerve tube in addition. Clinical Follow-up will be performed after 3,6,12 and 24 months.
  Arms: Chitosan
Procedure: Gold standard Primary microsurgical repair — Primary microsurgical repair of traumatic lesion of sensory nerves of the hand. Clinical Follow-up will be performed after 3,6,12 and 24 months.

SUMMARY:
The objective of this study is to evaluate whether the additional use of a nerve tube in primary microsurgical repair of traumatic sensory nerve lesions of the hand has an effect on convalescence and functional results.

DETAILED DESCRIPTION:
Standard therapy for nerve injuries of the hand without a gap is a direct tension free microsurgical repair. Often, a nerve tube is used in addition to a direct nerve suture to protect the nerve from scar formation and guide the regenerating axons to the distal stump, but there is still a lack of data for this approach. The basic design of these nerve tubes is similar but they are made of different resorbable biomaterials. Chitosan, a derivative of chitin, is biocompatible and is similar to natural glycosaminoglycans. In vivo studies showed positive effects on the survival and orientation of Schwann cells as well as the survival and differentiation of neuronal cells and prevention of painful neuromas. Therefore it is the ideal material for a nerve tube. In this study we want to test a Chitosan based nerve tube (already certified German medical product with European label (CE-label)) - as an additional treatment for digital nerve injuries without a gap.

This study will enroll participants with traumatic sensory nerve lesions from 3 Centres: Trauma Center Ludwigshafen (Ludwigshafen, Germany), Trauma Center Frankfurt am Main (Frankfurt am Main, Germany) and Trauma Center Bochum (Bochum, Germany). After being informed about the study and its potential risks, patients with traumatic sensory nerve lesions will be consecutively screened for eligibility. The study will be conducted in four successive periods. All enrolled participants will be randomized locally by alternating local lists in the Double-Blind Period. After enrolment, the assigned subject number will be used on all Case Report Forms. The kind of intervention is blinded for the participant and for the investigator of the follow-up that was not involved in surgery. Enrolled participants will be randomized in a 1:1 ratio to primary microsurgical repair with the additional use of a nerve tube, or direct tension free microsurgical repair alone.

Data will be collected in Case Report Forms (CRFs) according to European DIN standard (International Standards Organization (EN ISO) 14155) and Good Clinical Practice recommendations. CRFs will be transmitted electronically to the executive study centre in Ludwigshafen and will be checked there for integrity, quality and consistency. The executive study centre will also ensure standardisation of the registry process, operative procedure and follow-up in all participating centers by periodic monitoring. Furthermore written instructions and a course of instruction will be provided to each Investigator. Data will be collected and analyzed in the executive study centre. There will be also CRFs for reporting drop-outs and for reporting adverse events.

The static 2-point-discrimination (2PD) after 6 months will bet the primary outcome parameter. Assumptions for the gold standard treatment can be made from literature. The mean of 2-PD after 6 months is approximately 8 mm with a standard deviation of 3 mm. A decrease of 2 mm in the 2-PD would be clinically relevant and is assumed for the experimental intervention. Using a 2-sided t-test with a level of 0.05 and a power of 80%, will require 37 patients per group in order to show superiority. The primary endpoint is tested in the per-protocol set (PPS) via an analysis of covariance with centre as factor and distance between lesion and finger pulp as covariate. Secondary objectives will be described without confirmatory analysis. In order to compensate a loss of follow-up or data 50 patients per group will be randomized.

ELIGIBILITY:
Inclusion Criteria:

* Primary complete traumatic lesion of sensory-only nerves of the hand without a defect zone
* Patient age between 18 an 67 years
* Informed Consent.

Exclusion Criteria:

* Amputated or avascular fingers
* Known impaired sensibility of the injured finger
* Allergy to chitosan
* Pregnancy
* Immunodeficiency

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-03; Primary Completion 2017-07 (Actual); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Ability for two-point discrimination of the injured finger (2PD) (measured with compasses0 | 6 months after intervention
  The ability for static two-point discrimination of the injured finger will be measured with compasses in the 6 month follow-up.

SECONDARY OUTCOMES:
Ability for two-point discrimination of the injured finger (2PD) / Sensibility (checking patients ability to recognize filaments of different calibers.) | 3,6,12,24 months after intervention
  The ability for static two-point discrimination of the injured finger will be measured with compasses also in the other follow-ups. Furthermore, sensibility of the injured finger will be measured by
DASH-score | 3,6,12,24 months after intervention
  Patient's individual disability in activities of daily living will be measured with the DASH-questionnaire.
Grip strength | 3,6,12,24 months after intervention
  Grip strength of both hands will be measured with a dynamometer and will be compared to the opposite side.
Range of motion of the injured finger | 3,6,12,24 months after intervention
  The Range of motion of the injured finger will be measured with a goniometer for small joints and will be compared to the opposite side.
Pain (visual analogue scales) | 3,6,12,24 months after intervention
  Patients will self report pain on visual analogue scales, ranged from 0 (no pain) up to 10 (maximum of pain)
Cold intolerance (Grades: 0 = Hinders function; 1 = Disturbing; 2 = Moderate; 3 = None/minor) | 3,6,12,24 months after intervention
  The examiner will question the patient about cold intolerance. (Grades: 0 = Hinders function; 1 = Disturbing; 2 = Moderate; 3 = None/minor)
Hypersensitivity (Grades: 0 = Hinders function; 1 = Disturbing; 2 = Moderate; 3 = None/minor) | 3,6,12,24 months after intervention
  The examiner will stroke the dysfunctional area and question the patient about cold hypersensitivity. (Grades: 0 = Hinders function; 1 = Disturbing; 2 = Moderate; 3 = None/minor)
Existence of neuromas | 3,6,12,24 months after intervention
  The existence of a neuroma will be assessed clinically and by neurosonography.

OTHER OUTCOMES:
Adverse events | Participants will be followed for the duration of hospital stay, an expected average of 5 days and 3,6,12,24 months after intervention.
  Record of any type of revision surgery. Registration of the incidence of postoperative hematoma, deep wound infections, disturbances of scar formation.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Kremer, MD, Study Chair — BG Unfallklinik Ludwigshafen
Locations (3):
- Germany (3):
  - BG Universitätsklinikum Bergmannsheil Bochum, Bochum
  - BG Unfallklinik Frankfurt, Frankfurt
  - BG Unfallklinik Ludwigshafen, Ludwigshafen

REFERENCES:
- [Background] Ao Q, Fung CK, Tsui AY, Cai S, Zuo HC, Chan YS, Shum DK. The regeneration of transected sciatic nerves of adult rats using chitosan nerve conduits seeded with bone marrow stromal cell-derived Schwann cells. Biomaterials. 2011 Jan;32(3):787-96. doi: 10.1016/j.biomaterials.2010.09.046. Epub 2010 Oct 14. PMID 20950852
- [Background] Bowsher D. Human "autotomy". Pain. 2002 Jan;95(1-2):187-9. doi: 10.1016/s0304-3959(01)00389-x. PMID 11790481
- [Background] Chaise F, Friol JP, Gaisne E. [Results of emergency repair of wounds of palmar collateral nerves of the fingers]. Rev Chir Orthop Reparatrice Appar Mot. 1993;79(5):393-7. French. PMID 8066288
- [Background] Freier T, Koh HS, Kazazian K, Shoichet MS. Controlling cell adhesion and degradation of chitosan films by N-acetylation. Biomaterials. 2005 Oct;26(29):5872-8. doi: 10.1016/j.biomaterials.2005.02.033. Epub 2005 Apr 9. PMID 15949553
- [Background] Haastert-Talini K, Geuna S, Dahlin LB, Meyer C, Stenberg L, Freier T, Heimann C, Barwig C, Pinto LF, Raimondo S, Gambarotta G, Samy SR, Sousa N, Salgado AJ, Ratzka A, Wrobel S, Grothe C. Chitosan tubes of varying degrees of acetylation for bridging peripheral nerve defects. Biomaterials. 2013 Dec;34(38):9886-904. doi: 10.1016/j.biomaterials.2013.08.074. Epub 2013 Sep 17. PMID 24050875
- [Background] Hudak PL, Amadio PC, Bombardier C. Development of an upper extremity outcome measure: the DASH (disabilities of the arm, shoulder and hand) [corrected]. The Upper Extremity Collaborative Group (UECG). Am J Ind Med. 1996 Jun;29(6):602-8. doi: 10.1002/(SICI)1097-0274(199606)29:63.0.CO;2-L. PMID 8773720
- [Background] Kim DH, Han K, Tiel RL, Murovic JA, Kline DG. Surgical outcomes of 654 ulnar nerve lesions. J Neurosurg. 2003 May;98(5):993-1004. doi: 10.3171/jns.2003.98.5.0993. PMID 12744359
- [Background] Konofaos P, Ver Halen JP. Nerve repair by means of tubulization: past, present, future. J Reconstr Microsurg. 2013 Mar;29(3):149-64. doi: 10.1055/s-0032-1333316. Epub 2013 Jan 9. PMID 23303520
- [Background] Lewin-Kowalik J, Marcol W, Kotulska K, Mandera M, Klimczak A. Prevention and management of painful neuroma. Neurol Med Chir (Tokyo). 2006 Feb;46(2):62-7; discussion 67-8. doi: 10.2176/nmc.46.62. PMID 16498214
- [Background] Marcol W, Larysz-Brysz M, Kucharska M, Niekraszewicz A, Slusarczyk W, Kotulska K, Wlaszczuk P, Wlaszczuk A, Jedrzejowska-Szypulka H, Lewin-Kowalik J. Reduction of post-traumatic neuroma and epineural scar formation in rat sciatic nerve by application of microcrystallic chitosan. Microsurgery. 2011 Nov;31(8):642-9. doi: 10.1002/micr.20945. Epub 2011 Oct 18. PMID 22009638
- [Background] Meek MF, Coert JH. Recovery of two-point discrimination function after digital nerve repair in the hand using resorbable FDA- and CE-approved nerve conduits. J Plast Reconstr Aesthet Surg. 2013 Oct;66(10):1307-15. doi: 10.1016/j.bjps.2013.04.058. Epub 2013 Jul 2. PMID 23827446
- [Background] Scott J, Huskisson EC. Vertical or horizontal visual analogue scales. Ann Rheum Dis. 1979 Dec;38(6):560. doi: 10.1136/ard.38.6.560. PMID 317239
- [Background] Simoes MJ, Gartner A, Shirosaki Y, Gil da Costa RM, Cortez PP, Gartner F, Santos JD, Lopes MA, Geuna S, Varejao AS, Mauricio AC. In vitro and in vivo chitosan membranes testing for peripheral nerve reconstruction. Acta Med Port. 2011 Jan-Feb;24(1):43-52. Epub 2011 Feb 28. PMID 21672441
- [Background] Weber RA, Breidenbach WC, Brown RE, Jabaley ME, Mass DP. A randomized prospective study of polyglycolic acid conduits for digital nerve reconstruction in humans. Plast Reconstr Surg. 2000 Oct;106(5):1036-45; discussion 1046-8. doi: 10.1097/00006534-200010000-00013. PMID 11039375
- [Background] Xu H, Yan Y, Li S. PDLLA/chondroitin sulfate/chitosan/NGF conduits for peripheral nerve regeneration. Biomaterials. 2011 Jul;32(20):4506-16. doi: 10.1016/j.biomaterials.2011.02.023. Epub 2011 Mar 11. PMID 21397324
- [Background] Yuan Y, Zhang P, Yang Y, Wang X, Gu X. The interaction of Schwann cells with chitosan membranes and fibers in vitro. Biomaterials. 2004 Aug;25(18):4273-8. doi: 10.1016/j.biomaterials.2003.11.029. PMID 15046917
- [Background] Zimmermann M. Pathobiology of neuropathic pain. Eur J Pharmacol. 2001 Oct 19;429(1-3):23-37. doi: 10.1016/s0014-2999(01)01303-6. PMID 11698024
- [Derived] Neubrech F, Sauerbier M, Moll W, Seegmuller J, Heider S, Harhaus L, Bickert B, Kneser U, Kremer T. Enhancing the Outcome of Traumatic Sensory Nerve Lesions of the Hand by Additional Use of a Chitosan Nerve Tube in Primary Nerve Repair: A Randomized Controlled Bicentric Trial. Plast Reconstr Surg. 2018 Aug;142(2):415-424. doi: 10.1097/PRS.0000000000004574. PMID 30045179
- [Derived] Neubrech F, Heider S, Harhaus L, Bickert B, Kneser U, Kremer T. Chitosan nerve tube for primary repair of traumatic sensory nerve lesions of the hand without a gap: study protocol for a randomized controlled trial. Trials. 2016 Jan 26;17:48. doi: 10.1186/s13063-015-1148-5. PMID 26811067